CLINICAL TRIAL: NCT04946019
Title: A Prospective, Phase II Study of MR-Linac Guided Adaptive Fractionated Stereotactic Radiotherapy for Brain Metastases From Non-small Cell Lung Cancer
Brief Title: MR-Linac Guided Adaptive FSRT for Brain Metastases From Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1075
Record Dates: First submitted 2021-06-25; First posted 2021-06-30 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; MR-Linac; Fractionated stereotactic radiation therapy; Brain metastase
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-Linac Guided Adaptive FSRT (Experimental): Patients will receive FSRT (30Gy in 5 fractions) on the MR-Linac treatment machine.
  Interventions: Combination Product: Unity-based MR-Linac guided FSRT

INTERVENTIONS:
Combination Product: Unity-based MR-Linac guided FSRT — The FSRT was delivered using the Unity-based MR-Linac treatment machine, with a total dose of 30Gy in 5 fractions.

SUMMARY:
This Phase II study is to determine the efficacy and safety of MR-Linac Guided Adaptive fractionated stereotactic radiotherapy (FSRT) in patients with brain metastases in non-small cell lung cancer.

DETAILED DESCRIPTION:
This Phase II study is to determine the efficacy and safety of MR-Linac Guided Adaptive fractionated stereotactic radiotherapy (FSRT) in patients with brain metastases in non-small cell lung cancer.

Patients will receive FSRT (30Gy in 5 fractions) on the MR-Linac treatment machine. The primary end point is 1-year intracranial progression-free survival. The secondary end points are objective response rate, 1-y PFS, 1-y OS, perilesional edema of brain metastases, quality of life, safety of treatment, dose coverage of targets and dose to normal organs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* Histologically or cytologically confirmed non-small cell lung cancer
* 1-10 metastases on contrast-enhanced MRI
* Radiotherapy for extracranial lesions is permitted
* Tyrosine kinase inhibitors (TKI) are permitted in patients with progression of intracranial metastases during previous TKI therapy
* Patients have measurable or evaluable lesions based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Normal function of organs and bone marrow within 14 days: Total bilirubin 1.5 times or less the upper limits of normal (ULN); AST and ALT 1.5 times or less the ULN; absolute neutrophil count≥ 500 cells/mm3; creatinine clearance rate(CCR) ≥45 mL/min; Platelet count≥50,000 cells/mm3; international normalized ratio(INR) ≤1.5#Prothrombin Time (PT)≤ 1.5 × ULN
* Informed-consent

Exclusion Criteria:

* Small cell carcinoma of lung
* Intracranial metastases needed surgical decompression
* Patients with contraindications for MRI
* Previous radiotherapy or excision for intracranial metastases
* The tumor has completely approached, encircled, or invaded the intravascular space of the great vessels (e.g., the pulmonary artery or the superior vena cava)
* A cavity over 2cm in diameter of primary tumor or metastasis
* Bleeding tendency or coagulation disorder
* Hemoptysis (1/2 teaspoon blood/day) happened within 1 month
* The use of full-dose anticoagulation within the past 1 month
* Severe vascular disease occurred within 6 months
* Gastrointestinal fistula, perforation or abdominal abscess occurred within 6 months
* Hypertensive crisis, hypertensive encephalopathy, symptomatic heart failure (New York class II or above), active cerebrovascular disease or cardiovascular disease occurred within 6 months
* Uncontrolled hypertension (systolic > 150mmHg and/or diastolic > 100mmHg)
* Major surgery within 28 days or minor surgery or needle biopsy within 48 hours
* Urine protein 3-4+, or 24h urine protein quantitative >1g
* Severe uncontrolled disease
* Uncontrollable seizure or psychotic patients without self-control ability
* Women in pregnancy, lactation period
* Other not suitable conditions determined by the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
1-year intracranial progression-free survival | 1 year

SECONDARY OUTCOMES:
Objective response rate | 2 months
1-year progression-free survival | 1 year
1-year overall survival | 1 year
Rate of participants with perilesional edema of brain metastases evaluated byT2-weighted MRI | 1 year
Quality of life evaluated by EORTC quality of life questionnaire | 1 year
Rate of patients with treatment-related adverse events evaluated by CTCAE v4.0 | 1 year
Dose coverage to targets | 2 months
Dose to normal organs | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Hui Liu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaw MG, Ball DL. Treatment of brain metastases in lung cancer: strategies to avoid/reduce late complications of whole brain radiation therapy. Curr Treat Options Oncol. 2013 Dec;14(4):553-67. doi: 10.1007/s11864-013-0258-0. PMID 24048959
- [Background] Yamamoto M, Serizawa T, Shuto T, Akabane A, Higuchi Y, Kawagishi J, Yamanaka K, Sato Y, Jokura H, Yomo S, Nagano O, Kenai H, Moriki A, Suzuki S, Kida Y, Iwai Y, Hayashi M, Onishi H, Gondo M, Sato M, Akimitsu T, Kubo K, Kikuchi Y, Shibasaki T, Goto T, Takanashi M, Mori Y, Takakura K, Saeki N, Kunieda E, Aoyama H, Momoshima S, Tsuchiya K. Stereotactic radiosurgery for patients with multiple brain metastases (JLGK0901): a multi-institutional prospective observational study. Lancet Oncol. 2014 Apr;15(4):387-95. doi: 10.1016/S1470-2045(14)70061-0. Epub 2014 Mar 10. PMID 24621620
- [Background] Rades D, Janssen S, Dziggel L, Blanck O, Bajrovic A, Veninga T, Schild SE. A matched-pair study comparing whole-brain irradiation alone to radiosurgery or fractionated stereotactic radiotherapy alone in patients irradiated for up to three brain metastases. BMC Cancer. 2017 Jan 6;17(1):30. doi: 10.1186/s12885-016-2989-3. PMID 28061768
- [Background] Baliga S, Garg MK, Fox J, Kalnicki S, Lasala PA, Welch MR, Tome WA, Ohri N. Fractionated stereotactic radiation therapy for brain metastases: a systematic review with tumour control probability modelling. Br J Radiol. 2017 Feb;90(1070):20160666. doi: 10.1259/bjr.20160666. Epub 2016 Dec 12. PMID 27936894
- [Background] Barrett OC, McDonald AM, Thompson JW, Bredel M, McGwin G, Riley KO, Fiveash JB. Distant brain recurrence in patients with five or more newly diagnosed brain metastases treated with focal stereotactic radiotherapy alone. J Radiosurg SBRT. 2017;4(4):255-263. PMID 28626600
- [Background] Lagendijk JJ, Raaymakers BW, Van den Berg CA, Moerland MA, Philippens ME, van Vulpen M. MR guidance in radiotherapy. Phys Med Biol. 2014 Nov 7;59(21):R349-69. doi: 10.1088/0031-9155/59/21/R349. Epub 2014 Oct 16. No abstract available. PMID 25322150
- [Background] MacManus M, Everitt S, Schimek-Jasch T, Li XA, Nestle U, Kong FS. Anatomic, functional and molecular imaging in lung cancer precision radiation therapy: treatment response assessment and radiation therapy personalization. Transl Lung Cancer Res. 2017 Dec;6(6):670-688. doi: 10.21037/tlcr.2017.09.05. PMID 29218270
- [Background] Khoo VS, Joon DL. New developments in MRI for target volume delineation in radiotherapy. Br J Radiol. 2006 Sep;79 Spec No 1:S2-15. doi: 10.1259/bjr/41321492. PMID 16980682
- [Background] Raaymakers BW, Lagendijk JJ, Overweg J, Kok JG, Raaijmakers AJ, Kerkhof EM, van der Put RW, Meijsing I, Crijns SP, Benedosso F, van Vulpen M, de Graaff CH, Allen J, Brown KJ. Integrating a 1.5 T MRI scanner with a 6 MV accelerator: proof of concept. Phys Med Biol. 2009 Jun 21;54(12):N229-37. doi: 10.1088/0031-9155/54/12/N01. Epub 2009 May 19. PMID 19451689
- [Background] Stemkens B, Tijssen RH, de Senneville BD, Lagendijk JJ, van den Berg CA. Image-driven, model-based 3D abdominal motion estimation for MR-guided radiotherapy. Phys Med Biol. 2016 Jul 21;61(14):5335-55. doi: 10.1088/0031-9155/61/14/5335. Epub 2016 Jun 30. PMID 27362636
- [Background] Dietz B, Yip E, Yun J, Fallone BG, Wachowicz K. Real-time dynamic MR image reconstruction using compressed sensing and principal component analysis (CS-PCA): Demonstration in lung tumor tracking. Med Phys. 2017 Aug;44(8):3978-3989. doi: 10.1002/mp.12354. Epub 2017 Jun 28. PMID 28543069
- [Background] Glitzner M, Crijns SP, de Senneville BD, Kontaxis C, Prins FM, Lagendijk JJ, Raaymakers BW. On-line MR imaging for dose validation of abdominal radiotherapy. Phys Med Biol. 2015 Nov 21;60(22):8869-83. doi: 10.1088/0031-9155/60/22/8869. Epub 2015 Nov 4. PMID 26531846
- [Background] Kontaxis C, Bol GH, Stemkens B, Glitzner M, Prins FM, Kerkmeijer LGW, Lagendijk JJW, Raaymakers BW. Towards fast online intrafraction replanning for free-breathing stereotactic body radiation therapy with the MR-linac. Phys Med Biol. 2017 Aug 21;62(18):7233-7248. doi: 10.1088/1361-6560/aa82ae. PMID 28749375
- [Background] Raaymakers BW, Jurgenliemk-Schulz IM, Bol GH, Glitzner M, Kotte ANTJ, van Asselen B, de Boer JCJ, Bluemink JJ, Hackett SL, Moerland MA, Woodings SJ, Wolthaus JWH, van Zijp HM, Philippens MEP, Tijssen R, Kok JGM, de Groot-van Breugel EN, Kiekebosch I, Meijers LTC, Nomden CN, Sikkes GG, Doornaert PAH, Eppinga WSC, Kasperts N, Kerkmeijer LGW, Tersteeg JHA, Brown KJ, Pais B, Woodhead P, Lagendijk JJW. First patients treated with a 1.5 T MRI-Linac: clinical proof of concept of a high-precision, high-field MRI guided radiotherapy treatment. Phys Med Biol. 2017 Nov 14;62(23):L41-L50. doi: 10.1088/1361-6560/aa9517. PMID 29135471
- [Background] Ma LH, Li G, Zhang HW, Wang ZY, Dang J, Zhang S, Yao L, Zhang XM. Hypofractionated stereotactic radiotherapy with or without whole-brain radiotherapy for patients with newly diagnosed brain metastases from non-small cell lung cancer. J Neurosurg. 2012 Dec;117 Suppl:49-56. doi: 10.3171/2012.7.GKS121071. PMID 23205789
- [Derived] Zheng S, Ding S, Liu B, Xiong Y, Zhou R, Zhang P, Liu F, Liu Y, Chen M, Situ Y, Wang M, Huang X, Yin S, Fang W, Mou Y, Qiu B, Wang D, Liu H. Efficacy and safety of online adaptive magnetic resonance-guided fractionated stereotactic radiotherapy for brain metastases in non-small cell lung cancer (GASTO-1075): a single-arm, phase 2 trial. EClinicalMedicine. 2025 Apr 9;82:103189. doi: 10.1016/j.eclinm.2025.103189. eCollection 2025 Apr. PMID 40247887